CLINICAL TRIAL: NCT03619161
Title: Bleach vs. Bubbles: Assessing the Impact of the Bathroom Environment on Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1227
Record Dates: First submitted 2018-07-27; First posted 2018-08-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Eczema; Atopic Dermatitis; Atopic Dermatitis and Related Conditions
Keywords: atopic dermatitis; eczema; bleach bath; bacteria; bathroom; cleaning
MeSH Terms: conditions — Eczema; Dermatitis, Atopic | interventions — Gastric Balloon

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No cleaning (control) (No Intervention): Patients will have a bacterial culture taken from their bathtub and then continue regular care. We will offer to clean their bathrooms after the 4 week intervention period ends.
- Bubbles (Experimental): Patients will have a bacterial culture taken from their bathtub and have their bathrooms cleaned by the investigators
  Interventions: Other: Bubbles
- Bleach and Bubbles (Active Comparator): Patients will have a bacterial culture taken from their bathtub, have their bathrooms cleaned by the investigators, and be given instructions to perform bleach baths twice weekly.
  Interventions: Other: Bleach and Bubbles

INTERVENTIONS:
Other: Bubbles — All bathrooms with showers or bathtubs will be cleansed with simple products (dilute bleach, dilute white vinegar, baking soda, and dilute Dawn dish soap)
  Other Names: cleaning
  Arms: Bubbles
Other: Bleach and Bubbles — All bathrooms with showers or bathtubs will be cleansed with simple products (dilute bleach, dilute white vinegar, baking soda, and dilute Dawn dish soap).
  Other Names: cleaning; bleach bath
  Arms: Bleach and Bubbles

SUMMARY:
Purpose: Evaluate the impact of cleaning the bathroom environment on the severity of eczema. Determine if part of the efficacy of bleach baths may be in cleaning the bathroom. Record data on the process in order to improve future interventions.

Participants: Patients and families with eczema

Procedures (methods):

* Obtain baseline eczema severity scores and bacterial cultures from bathtubs
* Randomize subjects to receive (1) a bathtub culture alone; (2) a culture and bathroom cleaning; and (3) a culture, cleaning, and bleach baths.
* Measure changes in eczema severity scores over 4 weeks
* Qualitatively evaluate the process by participants and investigators

DETAILED DESCRIPTION:
The study will evaluate the effect of two interventions.

1. At the start of the study, two-thirds of the patients (40 patients) will be randomized to have a culture taken from their bathtub with subsequent cleaning of all of their bathrooms (intervention arm) versus one-third (20 patients) only obtaining a culture taken from their bathtub with no cleaning (control arm).
2. After cleansing the bathrooms in the intervention arm, this group will be randomized again so that half of this group (20 patients) receives instructions on performing twice weekly bleach baths and the other half (20 patients) does not.
3. When the intervention period ends at 4 weeks, the placebo arm will be offered a bathroom cleaning.

There will be four quantitative assessment phases:

1. Upon entry into the study the investigators will obtain basic demographic information (insurer, age, race/ethnicity), a history of skin infections and allergic diseases, an eczema severity score (POEM score), an eczema area and severity index score (EASI score), and record the participant's level of eczema therapy (weak-moderate topical steroids, strong topical steroids, or systemic immunomodulators).
2. The investigators will obtain a culture from the bathtub used by every study subject. This will be prior to cleaning the bathroom if the participant is in the cleaning intervention arm.
3. The investigators will obtain a POEM score over the phone 1 week after obtaining the cultures.
4. After 4 weeks, the investigators will obtain a POEM score over the phone as well as document whether the participant received any antibiotics or had any visits to medical providers for atopy flares over the last 4 weeks. The investigators will also re-record the participant's level of eczema therapy (weak-moderate topical steroids, strong topical steroids, or systemic immunomodulators).

There will be one qualitative assessment:

Additionally, the study team will keep field notes documenting perceptions and experiences during the cleaning process. These qualitative documents will be used for process evaluation to improve home hygiene interventions and studies. Domains that the investigators will assess in field notes include:

1. Environment: The general appearance of the exterior of the home and neighborhood, cleanliness and order within the home and bathrooms, the hospitality and dynamics of interacting with the family. The investigators will also take pictures of the bathroom before and after each cleansing.
2. Work difficulty: Description of activities performed and any physical, mental, and emotional toil related to the labor with suggestions for improving the work experience.
3. Assessment of usefulness to the family: Did the family find the intervention useful? Did the family mention ways to make the cleaning intervention better? If given bleach bath instructions, did the family appear receptive and willing to do bleach baths? Did it appear that the family would clean their bathroom regularly after the intervention?

ELIGIBILITY:
Inclusion Criteria:

* Children with eczema who visit UNC pediatric dermatology during study enrollment (Summer 2018).
* Currently on a class 1 topical steroid or systemic immunosuppressive agent to control his/her eczema at the time of recruitment.
* A history of, or current clinical evaluation by the attending dermatologist showing, atopic dermatitis affecting at least 10% body surface area.

Exclusion Criteria:

* Child or family member with a sensitivity to bleach.
* Child has used bleach baths within the last 2 months.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Absolute change in POEM score From Baseline (day 0) to Week 4 (day 28) | Baseline (day 0) to Week 4 (day 28)
  POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease). A higher POEM score correlates with a poorer quality of life (QOL).

CONTACTS AND LOCATIONS:
Overall Officials: Craig N Burkhart, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share deidentified individual data that supports the results. This may include the study protocol, the statistical analysis plan, and/or the spreadsheet used to collect data.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available beginning 9 to 36 months following publication provided the investigator meets the appropriate access criteria.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.